CLINICAL TRIAL: NCT02922660
Title: Comparison of Desflurane Balanced Anesthesia Versus TIVA-TCI (Total IntraVenous Anesthesia-Target Controlled Infusion) in Patients Undergoing Ophthalmic Ambulatory Surgery: A Single Center, Prospective, Randomized, Controlled Study
Brief Title: Comparison of Desflurane Anesthesia Versus TIVA-TCI in Patients Undergoing Ophthalmic Ambulatory Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaoliang Gan (Other)
Responsible Party: Sponsor-Investigator, Xiaoliang Gan, associate chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ZOCMZK-2016
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Ophthalmic; Surgery; Anesthesia
Keywords: Ambulatory surgery; Ophthalmic; Inhalation anesthesia; Desflurane; Total intravenous anesthesia
MeSH Terms: interventions — Desflurane; Anesthesia, Inhalation; Propofol; Remifentanil; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group TIVA (Experimental): method of anesthesia is total intravenous anesthesia(TIVA) and maintenance with propofol Cp 2-4 μg/ml and remifentanil 2-4 ng/ml in target controlled infusion(TCI) during the procedure
  Interventions: Procedure: total intravenous anesthesia; Drug: Propofol; Drug: Remifentanil
- Group Des (Experimental): method of anesthesia is inhalation anesthesia and maintenance with desflurane ranged from 0.5~1.5 MAC during the procedure
  Interventions: Drug: desflurane; Procedure: inhalation anesthesia

INTERVENTIONS:
Drug: desflurane — method of anesthesia maintenance with desflurane ranged from 0.5~1.5 MAC during the procedure
  Other Names: Ethane,2--1,1,1,2-tetrafluoro
  Arms: Group Des
Procedure: total intravenous anesthesia — method of anesthesia in group TIVA is total intravenous anesthesia(TIVA) during the procedure
  Other Names: TIVA
  Arms: Group TIVA
Procedure: inhalation anesthesia — method of anesthesia in group DES is inhalation anesthesia with desflurane during the procedure
  Arms: Group Des
Drug: Propofol — using propofol as sedative during the procedure of anesthesia and maintaining with propofol Cp 2-4 μg/ml in TCI
  Other Names: Disoprofol
  Arms: Group TIVA
Drug: Remifentanil — using remifentanil as analgesics during the procedure of anesthesia and maintaining with remifentanil 2-4 ng/ml in TCI
  Other Names: Remifentanil Hydrochloride for Injection
  Arms: Group TIVA

SUMMARY:
This is a single-center, randomized, prospective research which aims to investigate the advantages and disadvantages between desflurane balanced anesthesia and TIVA-TCI with propofol in ophthalmic ambulatory surgery, so that to evaluate a better anesthesia method in ophthalmic surgery through a large sample clinical study.

DETAILED DESCRIPTION:
Desflurane balanced anesthesia and TIVA-TCI(Total IntraVenous Anesthesia-Target Controlled Infusion) are commonly used in ophthalmic ambulatory surgery, however, there is no clear evidence to discriminate the advantages and disadvantages between them. This study is designed to evaluate a better anesthetic method in ophthalmic surgery through a clinical study. This is a single center, randomized, prospective study. 200 patients with American Society of Anesthesiologists'(ASA) physical status 1 to 2, aged 18 to 60, scheduled for elective strabismus ambulatory and in whom a LMA is indicated for anesthesia are recruited. Enrolled patients are randomly assigned into 2 groups: group TIVA (TIVA-TCI with propofol) and group Des (Desflurane).In group TIVA, anesthesia is maintained with propofol and remifentanil. Propofol is continuously administered via a target-controlled infusion (TCI) pump intraoperatively. In group Des, anesthesia is maintained with desflurane.All patients received anaesthesia depth monitoring with bispectral index (BIS). The dose of anesthetic is adjusted to maintained the BIS value within 40 to 60. At the end of the surgery, inhalant anesthetic or infused propofol and remifentanil are discontinued. LMA is removed when patient regains consciousness with spontaneous respiration. Patients are then transferred to the post anesthetic care unit (PACU) for postoperative follow-up. The primary outcome is awake time, the secondary outcomes include discharge time, the stay time in PACU, time of off-bed, Riker sedation agitation score (SAS), time of PADSS>9, NRS score when leaving PACU, incidence of various complications (postoperative nausea and vomiting (PONV), emergence agitation, etc), as well as anesthesia cost. All patients are followed up by calling in one day after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years patients undergoing selective ophthalmic ambulatory surgery；
* ASA I and II
* duration of anesthesia at least 30min
* without apparent organ comorbidities
* sign the informed consent form

Exclusion Criteria:

* equal or greater than ASA III
* has a history of dementia，psychiatric disorders or central nervous system diseases
* taking sedatives, antidepressant or glucocorticoid
* without family members
* has cardiac, respiratory，liver，kidney comorbidities
* uncontrolled hypertension（>180/100mmHg）
* laryngeal mask fail to insert, and change to tracheal intubation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Awake time | From the ending time of anesthesia until the recovery time of patient's consciousness, assessed up to half an hour postoperatively.
  "Anesthesia ends" means stop infusing or inhaling any anaesthetic.

SECONDARY OUTCOMES:
Discharge time | From the ending time of anesthesia until the time of extubation, assessed up to half an hour postoperatively.
  The standards of extubation are tidal volume(VT) 6～8 ml/kg，respiratory rate(RR) 10～12 times per minute，end-tidal carbon dioxide (ETCO2) 35～45 mmHg.
Stay time in the postoperative care unit | Measuring the stay time in postoperative care unit, assessed up to one hour postoperatively.
Quality of recovery in 1 day postoperatively | Start scaling when 1 day(24 hour) postoperatively.
  It will use telephone follow-up for the patients enrolled.
Incidences in postoperative nausea and vomiting(PONV) | Start scaling in 1 day(24 hour) postoperatively.
Incidences in postoperative agitation | Start scaling in 1 day(24 hour) postoperatively.
Anesthesia cost | During the procedure of anesthesia.
Postoperative VAS pain score | Start scaling in half an hour postoperatively when patient's consciousness returns.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan ophthalmic center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aylin P, Williams S, Jarman B, Bottle A. Trends in day surgery rates. BMJ. 2005 Oct 8;331(7520):803. doi: 10.1136/bmj.331.7520.803. No abstract available. PMID 16210281
- [Background] Neel ST. Effect of Conversion to Immediate Sequential Cataract Surgery on Ambulatory Surgery Centers in the United States in the Cost-Analysis Model. JAMA Ophthalmol. 2015 Jul;133(7):856-7. doi: 10.1001/jamaophthalmol.2015.0941. No abstract available. PMID 25906175
- [Background] Chen CH, Yang YL, Chen WM, Shyr MH. Comparison of the anesthesia profiles between sevoflurane-nitrous oxide and propofol-nitrous oxide conveyed by laryngeal mask airway in patients undergoing ambulatory gynecological surgery. Acta Anaesthesiol Taiwan. 2006 Jun;44(2):101-7. PMID 16845915
- [Background] Kumar G, Stendall C, Mistry R, Gurusamy K, Walker D. A comparison of total intravenous anaesthesia using propofol with sevoflurane or desflurane in ambulatory surgery: systematic review and meta-analysis. Anaesthesia. 2014 Oct;69(10):1138-50. doi: 10.1111/anae.12713. Epub 2014 May 22. PMID 24847783
- [Background] Coskun D, Celebi H, Karaca G, Karabiyik L. Remifentanil versus fentanyl compared in a target-controlled infusion of propofol anesthesia: quality of anesthesia and recovery profile. J Anesth. 2010 Jun;24(3):373-9. doi: 10.1007/s00540-010-0898-1. Epub 2010 Mar 13. PMID 20229001
- [Background] Majholm B, Bartholdy J, Clausen HV, Virkus RA, Engbaek J, Moller AM. Comparison between local anaesthesia with remifentanil and total intravenous anaesthesia for operative hysteroscopic procedures in day surgery. Br J Anaesth. 2012 Feb;108(2):245-53. doi: 10.1093/bja/aer337. Epub 2011 Nov 23. PMID 22113931
- [Background] Eikaas H, Raeder J. Total intravenous anaesthesia techniques for ambulatory surgery. Curr Opin Anaesthesiol. 2009 Dec;22(6):725-9. doi: 10.1097/ACO.0b013e3283310f6b. PMID 19680121
- [Background] Yoo YC, Bai SJ, Lee KY, Shin S, Choi EK, Lee JW. Total intravenous anesthesia with propofol reduces postoperative nausea and vomiting in patients undergoing robot-assisted laparoscopic radical prostatectomy: a prospective randomized trial. Yonsei Med J. 2012 Nov 1;53(6):1197-202. doi: 10.3349/ymj.2012.53.6.1197. PMID 23074122
- [Background] Rinehardt EK, Sivarajan M. Costs and wastes in anesthesia care. Curr Opin Anaesthesiol. 2012 Apr;25(2):221-5. doi: 10.1097/ACO.0b013e32834f00ec. PMID 22157199
- [Derived] Zhu YL, Shen WH, Chen QR, Ye HJ, Huang JX, Kang Y, Chi W, Gan XL. Desflurane anesthesia compared with total intravenous anesthesia on anesthesia-controlled operating room time in ambulatory surgery following strabotomy: a randomized controlled study. Chin Med J (Engl). 2020 Apr 5;133(7):779-785. doi: 10.1097/CM9.0000000000000728. PMID 32149764